CLINICAL TRIAL: NCT04856566
Title: Examine the Feasibility of a Standardized Field Test for Marijuana and Alcohol Impairment: Laboratory Evaluations
Acronym: Alc-NHTSA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Highway Traffic Safety Administration (NHTSA) (U.S. Federal Agency); Hartford Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Godfrey Pearlson, Principal Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: HHC-2020-0368; DTNH2216C00022 (Other: Department of Transportation)
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-07

CONDITIONS: Marijuana Impairment; Alcohol Impairment
Keywords: marijuana; THC; cannabis; alcohol; driving
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols; Dronabinol; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low Dose THC + 0.05 BAC Alc (Experimental): Participants will receive low dose of THC along with alcohol leading to a BAC of 0.05.
  Interventions: Drug: Low Marijuana, Hash, THC, or Grass; Drug: 0.05 BAC Alcohol
- High Dose THC + 0.05 BAC Alc (Experimental): Participants will receive high dose of THC along with alcohol leading to a BAC of 0.05.
  Interventions: Drug: High Marijuana, Hash, THC, or Grass; Drug: 0.05 BAC Alcohol
- Placebo Drug + 0.05 BAC Alc (Experimental): Participants will receive placebo drug with no THC along with alcohol leading to a BAC of 0.05.
  Interventions: Drug: Placebo; Drug: 0.05 BAC Alcohol
- Placebo Drug + 0.08 BAC Alc (Experimental): Participants will receive placebo drug with no THC along with alcohol leading to a BAC of 0.08.
  Interventions: Drug: Placebo; Drug: 0.08 BAC Alcohol

INTERVENTIONS:
Drug: Low Marijuana, Hash, THC, or Grass — Cannabis with low amount of THC
  Other Names: Marijuana; THC
  Arms: Low Dose THC + 0.05 BAC Alc
Drug: High Marijuana, Hash, THC, or Grass — Cannabis with high amount of THC
  Other Names: Marijuana; THC
  Arms: High Dose THC + 0.05 BAC Alc
Drug: Placebo — Placebo drug with no THC
  Arms: Placebo Drug + 0.05 BAC Alc; Placebo Drug + 0.08 BAC Alc
Drug: 0.05 BAC Alcohol — Amount of alcohol when consumed leads to BAC of 0.05
  Arms: High Dose THC + 0.05 BAC Alc; Low Dose THC + 0.05 BAC Alc; Placebo Drug + 0.05 BAC Alc
Drug: 0.08 BAC Alcohol — Amount of alcohol when consumed leads to BAC of 0.08
  Arms: Placebo Drug + 0.08 BAC Alc

SUMMARY:
Alcohol and Cannabis (CNB) are two of the most widely used intoxicants. The effects of driving while intoxicated on alcohol are well documented, resulting in numerous drunken driving laws and regulations. As CNB begins to be decriminalized, medical CNB use allowed in multiple U.S. states, and perception of harmfulness falls, CNB use is predicted to rise and it will become increasingly common to publicly encounter persons who recently used the drug. An area of potentially high concern is if ever-greater numbers of CNB users and its legalization will increase the risk of driving while intoxicated from recent CNB use, thereby increasing the risks to public safety. This study aims to examine the combined effects of smoking marijuana and drinking alcohol on simulated driving.

DETAILED DESCRIPTION:
Alcohol is one of the most widely used substances. The effects of driving while intoxicated are well documented, leading to laws and regulations behind drunk driving. Marijuana is also a commonly abused drug. Marijuana use is not specific to social class, is linked to cognitive impairment and may be the cause of intoxication-induced accidents. The effects of marijuana intoxication on driving impairments are less documented. Data is being gathered in regards to this risk from our Neuroscience of Marijuana Impaired Driving study. The principle investigator's previous research includes the Brain and Alcohol Research with College Students (BARCS) study along with additional epidemiological studies reveal that most marijuana smokers also consume alcohol when they are intoxicated. These drugs interact pharmacodynamically and change each other's levels in the user's blood. They both have deleterious effects on driving. These effects are not additive but rather multiplicative. Someone using both substances will show more deleterious effects than someone using just one of these substances. This study will aim to investigate the brain and behavior in the same individuals, using a similar design to the NHTSA: Examine the Feasibility of a Standardized Field Test for Marijuana Impairment study. This structure coupled with past alcohol driving studies (Marijauna and Alcohol Impaired Driving) uses similar techniques of other measures of drunk driving. We hypothesize that alcohol and marijuana use combined will lead to greater impairment in a simulated driving task, as well as other driving related cognitive impairments. This study will aim to study feasible roadside sobriety tests for marijuana impairment.

The study will consist of 5 days (screening visit and 4 dose visit days). In a randomized, counterbalanced, double-blind study, investigators will dose participants with alcohol to a legal amount of 0.05% blood alcohol content on 3 study days and dose to 0.08% blood alcohol content on 1 study day. Then investigators will administer high THC marijuana, low THC marijuana or placebo marijuana using paced inhalation through a vaporizer. Participants will include 12 regular alcohol consumers aged 21 to 40 years of age; all participants must report smoking and drinking together. Following this dosing, investigators will assess impairment through cognitive testing as well as a simulated driving test and neuropsychological tests. Samples of blood will also be collected at multiple time points throughout the study visits to be measured for THC concentration and its metabolites. This allows clarification between the relationship of impairment, as well as subjective and objective intoxication, and levels of THC and it's metabolites in the users system.

ELIGIBILITY:
Inclusion Criteria:

* Must have a driver's license; recent 2 years highway driving experience
* Cannabis use for at least the past 2 years and report of getting high when smoking cannabis to avoid recruiting novice/inexperienced users.
* Reports regularly drinking and smoking (does not need to be at the same time)
* Use cannabis at least 5 times within life up to daily use, with occasional day of abstinence with no symptoms of craving or withdrawal.

Exclusion Criteria:

* Pregnancy, breastfeeding, and ineffective birth control methods.
* Current severe substance use disorder (except cannabis and tobacco substance use disorders)
* history of adverse effects with cannabis use
* serious medical, neuro-ophthalmological, or neurological illness (i.e. cancer, seizure disorders, encephalopathy)
* current diagnosis of any DSM-5 psychiatric disorder
* prior diagnosis of any DSM-5 psychiatric disorder
* report of any psychotic disorder in a first-degree relative
* history of head trauma with loss of consciousness > 30 minutes or concussion lasting 30 days.
* any medical/neurological condition that could compromise neurocognitive performance (i.e. epilepsy, multiple sclerosis, fetal alcohol syndrome)
* recovering alcoholics or anyone currently abstaining from alcohol.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Marijuana and alcohol induced performance changes on Cogstate 1-back/2-back task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Cogstate 1-back/2-back task assesses working memory, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on the Cogstate Social/Emotional Cognition Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Cogstate Social/Emotional Cognition task assesses emotional processing, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on Cogstate Card Learning. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Cogstate Card Learning task assesses visual memory, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on Groton Maze Learning task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Cogstate Groton Maze Learning task assesses spatial learning and memory, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on Alertmeter. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Alertmeter task assess visual judgment and alertness, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on the Time Estimation task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Time Estimation Task assesses timing, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on the Go-No-Go task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Go-No-Go task assesses inhibitory processing, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on the Ramaeker's Critical Tracking Test. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Raemaker's Critical Tracking Test assesses hand eye coordination and visuomotor tracking, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on the ANAM Pursuit Tracking Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The ANAM Pursuit Tracking Task assesses hand eye coordination, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on the Finger to Nose Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Finger to Nose Task assesses general motor coordination, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on the One Leg Stand Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The One Leg Stand Task assesses general motor coordination, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on the Line Walking/Months Backwards Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Line Walking/Months Backwards Task assesses general motor coordination plus distraction, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on the Time Reproduction Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  The Time Reproduction Task assesses general motor coordination plus timing, it will be administered prior to dosing and at various time points after dosing.
Marijuana and alcohol induced performance changes on the Ipod Balance Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  Participants will have an elastic wrap around their hips with an Ipod attached via durable velco. They will be asked to stand with both feet flat on the ground, looking ahead at a fixed point on the wall for 30 seconds, as well as 30 seconds with eyes closed. The amount of body sway will be measured using the accelerometer in an Ipod.
Marijuana and alcohol induced performance changes on the Ipod Punching Task. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  Participants will have an elastic wrap around their forearm with an Ipod attached via durable velrco. They will be asking to punch their arm forward while seated in a chair to measure their peak velocity of punching through the accelerometer in the Ipod.
Marijuana and alcohol induced performance changes on the DRUID tasks. | Baseline and post drug administration at: 10 min; 1.5 hours 2.5 hours
  DRUID is an application that has been designed to measure cognitive and behavior impairment following ingestion of drugs such as alcohol or marijuana. DRUID includes four Tasks to measure performance. The tasks are based on research on driving impairment and take about 5 minutes to complete. These tasks include a Reaction Time/Decision Making/DAT in which the subject has to press in two different locations on the Ipod screen dependent on which target shape appeared. The second task is a Reaction Time/Time Estimation/DAT task in which the subjects has to internally count up to 60 seconds while also touching the screen each time a target shape appears on the screen. The third task is a Motor Tracking/DAT tasks in which the subject must keep their finger on a moving circle on the screen. The last task is a balance task in which the subject is told to stand on one foot with the Ipod in an opposite hand keeping it as still as possible.

SECONDARY OUTCOMES:
Change in concentration of THC/metabolites in blood samples. | Baseline and post drug administration at: 30 min; 2.5 hours
  Blood samples with be collected at 3 times throughout each day to assess for changes of THC and its metabolite levels.
Change in concentration of THC/metabolites in oral fluid tested using Quantisal Oral Fluid Collection devices. | Baseline and post drug administration at: 30 min; 2.5 hours
  Oral fluid samples with be collected at 3 times throughout each day to assess for changes of THC and its metabolite levels.
Change in performance on simulated driving Road Tracking Task. | Post drug administration at: 30 min; 2.5 hours, 5 hours
  The Road Tracking Task measures operational control of the vehicle. Operational control is measured by standard deviation of lane position from the center point of the lane.
Change in performance on simulated driving Car Following Task. | Post drug administration at: 30 min; 2.5 hours, 5 hours
  The Car Following Task measures tactical control of the vehicle. Tactical control of the vehicle is measured by following distance from a lead vehicle.
Change in performance on simulated driving Gap Acceptance Task. | Post drug administration at: 30 min; 2.5 hours, 5 hours
  The Gap Acceptance Task measures strategic control of the vehicle. Strategic control of the vehicle is measured by size of headway gaps that the participant chooses in pulling out into oncoming traffic to overtake a stopped car.

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Pearlson, M.D, Principal Investigator — Founding Director, Olin Neuropsychiatry Center; Yale University
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States